CLINICAL TRIAL: NCT02119377
Title: A Mixed-Methods Study of Mental Health and Associated Factors in Transgender and Transsexual (Trans) People
Brief Title: First Australian National Trans Mental Health Study
Status: Completed | Type: Observational
Sponsor: Curtin University (Other)
Collaborators: Beyondblue (The National Depression Initiative) (Other)
Responsible Party: Principal Investigator, Zoë Hyde, Dr, Curtin University
Other Study IDs: CB:gc:6722
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Transsexualism
Keywords: trans; transsexual; transgender; sistergirl; brotherboy; androgynous; genderqueer
MeSH Terms: conditions — Transsexualism | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transgender and Transsexual People: Transgender and transsexual (trans) people aged 18 years or older living in Australia were invited to complete a questionnaire assessing a range of mental and physical health domains.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire

SUMMARY:
This is an Internet-based survey of transgender and transsexual (trans) people aged 18 years and older living in Australia. This population has received limited attention from public health researchers, planners, and practitioners. However, a growing body of evidence suggests that trans people experience disparities in several important areas of health compared with the population generally. In particular, trans people are more likely to experience mental health problems (notably depression and anxiety disorders), use alcohol, tobacco, and illicit drugs, and think about or attempt suicide. Additionally, trans people commonly report that their physical and mental health needs are not met, and underutilise preventive health care.

Participants were recruited using several non-probability sampling techniques, (including purposive sampling and snowball sampling), because random sampling is not possible with this population. Medical, social, support, and advocacy networks used by trans people were used to promote the study. A mixed quantitative and qualitative methodology was used. Validated quantitative instruments were used to obtain measures of health and well-being, which will be compared against population norms. Qualitative items complement these measures, providing rich experiential data.

The investigators hypothesised that:

* the prevalence of depressive and anxiety disorders will be higher than for the population generally, and that these conditions will commonly be undiagnosed and untreated;
* depressive and anxiety disorders will be associated with risky behaviours, such as tobacco, alcohol, and illicit drug use; and,
* trans people will report poor relationships with medical practitioners.

The investigators hypothesised that poor mental health is a consequence of several interrelated factors: body dysphoria (as a consequence of experiencing difficulty accessing medical treatment to alter sexual characteristics); societal discrimination and stigma (including harassment and violence); institutionalised discrimination (including difficulty changing identifying documents, and exclusion of surgical procedures and related treatments from public and private health systems); social isolation; and the belief held by many clinicians that transsexualism is a mental disorder (which may be a barrier to trans people forming trusting relationships with medical practitioners).

ELIGIBILITY:
Inclusion Criteria:

* Live in Australia
* Self-identify as trans

Exclusion Criteria:

* Aged less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a study of trans people living in Australia aged 18 years or older. The investigators used the term trans in an inclusive way, and included people who use (or used) words like transsexual, transgender, sistergirl, brotherboy, androgynous, or genderqueer to describe themselves. All trans people, including those who just describe themselves as men or women were encouraged to participate.
Sampling Method: Non-Probability Sample
Enrollment: 946 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of depressive and anxiety disorders | At time of entry into study (cross-sectional)
  Assessed by self-report, and with the Patient Health Questionnaire (PHQ)
Perceived physical and mental health status | At time of entry into study (cross-sectional)
  Assessed with the 36-item Short Form Health Survey (SF-36)

SECONDARY OUTCOMES:
Use of alcohol, tobacco, and illicit drugs | At time of entry into study (cross-sectional)
  Assessed by self-report
Patient-doctor relationship between trans people and their general practitioners, and doctors generally | At time of entry into study (cross-sectional)
  Assessed with the Patient-Doctor Relationship Questionnaire (PDRQ-9) and other quantitative and qualitative questions
Body image | At time of entry into study (cross-sectional)
  Assessed with the Body Image Quality of Life Inventory (BIQLI)
Factors that encourage and discourage trans people from accessing health care | At time of entry into study (cross-sectional)
  Assessed with qualitative questions
Factors that protect and promote mental health in trans people | At time of entry into study (cross-sectional)
  Assessed with qualitative questions
Use of hormone therapy and desire for, and uptake of transition-related surgery | At time of entry into study (cross-sectional)
  Assessed with quantitative and qualitative questions
Experiences of discrimination and harassment | At time of entry into study (cross-sectional)
  Assessed with quantitative and qualitative questions
Desire to, and success changing identifying documentation | At time of entry into study (cross-sectional)
  Assessed with quantitative and qualitative questions

CONTACTS AND LOCATIONS:
Overall Officials: Zoë Hyde, MPH PhD, Principal Investigator — Curtin University; Maryanne Doherty, MSc PhD, Principal Investigator — Curtin University; Peter Tilley, MPsych, Principal Investigator — Curtin University; Kieran A. McCaul, MPH PhD, Principal Investigator — The University of Western Australia; Rosanna Rooney, MPsych PhD, Principal Investigator — Curtin University; Jonine Jancey, PhD, Principal Investigator — Curtin University
Locations (1):
- Curtin University, Perth, Western Australia, Australia

REFERENCES:
- See also: Study website — http://transoz.org/